CLINICAL TRIAL: NCT02274428
Title: Phase 1 Clinical Trial of PNEUMOSTEM® Treatment in Premature Infants With Intraventricular Hemorrhage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Soon Park, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-06-103
Record Dates: First submitted 2014-10-02; First posted 2014-10-24 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Mesenchymal Stromal Cells
Keywords: intraventricular hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pneumostem group (Other): single arm, pneumostem treated infants
  Interventions: Drug: pneumostem

INTERVENTIONS:
Drug: pneumostem — human umbilical cord blood derived mesenchymal stem cells

SUMMARY:
Phase 1 clinical trial for the safety and dose determination of Pneumostem (human umbilical cord blood derived mesenchymal stem cells) in the premature infants with intraventricular hemorrhage (IVH, grade 3-4)

ELIGIBILITY:
Inclusion Criteria:

* 23-34w
* IVH grade 3-4, confirmed with brain ultrasonogram
* within 7 days after IVH diagnosis

Exclusion Criteria:

* severe congenital anomaly
* intrauterine intracranial bleeding
* intracranial infection
* severe congenital infection
* active and uncontrolled infection, CRP>10mg/dl
* Platelet count <50,000/ml
* severe metabolic acidosis (PH<7.1, BE<-20)

Ages: 23 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
unsuspected death or anaphylactic shock | within 6 h after pneumostem transplantation

SECONDARY OUTCOMES:
Death or hydrocephalus required shunt operation | First discharge home, maximum time frame : 1 year
  outcome measurement time frame would not exceed 1 year after birth

CONTACTS AND LOCATIONS:
Overall Officials: Won Soon Park, M.D. Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided